CLINICAL TRIAL: NCT03502434
Title: A Phase 1, Single-Center, Repeat Insult Patch Test (RIPT) Study Evaluating the Sensitization Potential of Topical SM04755 Solution
Brief Title: A Repeat Insult Patch Test (RIPT) Study Evaluating the Sensitization Potential of Topical SM04755 Solution in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SM04755-TOP-02
Record Dates: First submitted 2018-03-28; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Tendinopathy
MeSH Terms: conditions — Tendinopathy | interventions — Petrolatum; Sodium Dodecyl Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The Principal Investigator, subjects, and the site personnel who will be performing Reaction Grade assessments will be blinded to the Test Material identity, with the exception of the Positive Control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 90 mg/mL SM04755 in water (Experimental): 90 mg/mL SM04755 in water applied via patches
  Interventions: Drug: SM04755
- 90 mg/mL SM04755 in aqueous Vehicle (Experimental): 90 mg/mL SM04755 in aqueous Vehicle applied via patches
  Interventions: Drug: SM04755
- 90 mg/mL SM04755 in aqueous Vehicle (without Benzyl Alcohol) (Experimental): 90 mg/mL SM04755 in aqueous Vehicle (without Benzyl Alcohol) applied via patches
  Interventions: Drug: SM04755
- Vehicle (Other): Aqueous Vehicle applied via patches
  Interventions: Other: Vehicle
- White petrolatum (Other): White petrolatum (Negative control) applied via patches
  Interventions: Other: White Petrolatum
- Sodium lauryl sulfate (Other): Sodium lauryl sulfate (SLS 0.5%) (Positive control) applied via patches
  Interventions: Other: Sodium lauryl sulfate

INTERVENTIONS:
Drug: SM04755 — Healthcare professional-applied patches to subjects during the Induction Period on Days 1, 3, 5, 8, 10, 12, 15, 17 and 19, and during the Challenge Period on Day 36. Patches are to be worn by the subject for approximately 48-72 hours before removal and reaction grading.
  Arms: 90 mg/mL SM04755 in aqueous Vehicle; 90 mg/mL SM04755 in aqueous Vehicle (without Benzyl Alcohol); 90 mg/mL SM04755 in water
Other: Vehicle — Healthcare professional-applied patches to subjects during the Induction Period on Days 1, 3, 5, 8, 10, 12, 15, 17 and 19, and during the Challenge Period on Day 36. Patches are to be worn by the subject for approximately 48-72 hours before removal and reaction grading.
  Arms: Vehicle
Other: White Petrolatum — Healthcare professional-applied patches to subjects during the Induction Period on Days 1, 3, 5, 8, 10, 12, 15, 17 and 19, and during the Challenge Period on Day 36. Patches are to be worn by the subject for approximately 48-72 hours before removal and reaction grading.
  Arms: White petrolatum
Other: Sodium lauryl sulfate — Healthcare professional-applied patches to subjects during the Induction Period on Days 1, 3, 5, 8, 10, 12, 15, 17 and 19, and during the Challenge Period on Day 36. Patches are to be worn by the subject for approximately 48-72 hours before removal and reaction grading.
  Arms: Sodium lauryl sulfate

SUMMARY:
This is a single center, randomized, controlled, within subject comparison, single dose study to determine the sensitization potential of SM04755 solution on normal skin under semi-occlusive patch conditions.

DETAILED DESCRIPTION:
This Phase 1, Repeat Insult Patch Test (RIPT) study is a single-center study of topical SM04755 solution repetitively applied to skin of healthy volunteers. This study will assess the potential of the Test Materials to induce contact sensitization as measured by treatment emergent adverse events (TEAEs), Reaction Grade and Investigator assessment of irritation and sensitization.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and females at least 18 years of age
* Subjects of any Fitzpatrick skin type or race provided their degree of skin pigmentation does not, in the Investigator or designee's opinion, interfere with study assessments
* Subject has no signs of irritation (i.e., a Reaction Grade of "0") at patch application sites on the back prior to the initial patch application on Day 1
* Subject must have read, understood, and signed the informed consent form prior to any study-related procedure being performed
* Subject is willing and able to comply with all scheduled study visits, urine pregnancy tests (if applicable), contraception requirements (male and female), and other study requirements
* Subject is willing to avoid extensive sun exposure, phototherapy, or use of a tanning salon for the duration of the study

Exclusion Criteria:

* Women who are pregnant or lactating
* Women of childbearing potential who are sexually active and are not willing to use a highly effective method of birth control during the study period that includes double barrier, IUD, or hormonal contraceptive combined with single barrier, or abstinence
* Women of childbearing potential who have had unprotected sexual intercourse within 30 days prior to Day 1
* Males who are sexually active and not willing to use a condom, and have a partner who is capable of becoming pregnant, if neither has had surgery to become sterilized, and/or who are not willing to use double barrier or whose partner is not using a highly effective method of birth control (e.g., IUD, or hormonal contraception combined with single barrier)
* Subject has any skin condition that, in the Investigator's opinion, could interfere with the study assessments or put the subject at undue risk by study participation
* Subject has severe atopic dermatitis/eczema, psoriasis or chronic asthma
* Subject has tattoos, excessive hair, moles, scarring, etc. which would interfere with patching
* Subject has a history of sensitivity to any component of any of the Test Materials
* Use of any of the following medications:
* Systemic or topical glucocorticoids within 4 weeks prior to Day 1
* Systemic or topical analgesics (e.g., NSAIDs, high dose aspirin, etc.) within 1 week prior to Day 1. Note: Daily use of ≤325 mg of aspirin for cardiovascular disease or prophylaxis is allowed. Maximum daily use of Tylenol ≤3000 mg is allowed.
* Antihistamines within 1 week prior to Day 1. Note: H2 blockers such as Pepcid, Zantac, and Tagamet are permitted.
* Anti-inflammatories within 1 week prior to Day 1
* Immunosuppressant medications (e.g., TNF-alpha inhibitors, topical tacrolimus, etc.) within 4 weeks prior to Day 1 (or within 6 half-lives prior to Day 1 for biologics)
* Subject has had previous treatment with SM04755
* Subject has an active infection of hepatitis B or C or human immunodeficiency virus (HIV) infection as determined by an interview
* Participation in a clinical research trial that included the receipt of an investigational product or any experimental therapeutic procedure within 8 weeks prior to Screening, or planned participation in any such trial; the last date of participation in the trial, not the last date of receipt of investigational product, must be at least 8 weeks prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2017-11-17 (Actual)

PRIMARY OUTCOMES:
Contact sensitization potential of Test Material as measured by Treatment emergent | Baseline to Day 40 (or through the observation period for TEAEs)
Contact sensitization potential of Test Material as measured by Reaction Grade | Baseline to Day 38-40
  Reaction Grade is measured on a 5-point scale from zero to four (zero = no sign of irritation and 4 = Erythema with edema and blistering)
Contact sensitization potential of Test Material as measured by Investigator assessment of irritation and sensitization | Baseline to Day 40

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Yazici, M.D., Study Director — Biosplice Therapeutics, Inc.
Locations (1):
- Research Site, Lynchburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No